CLINICAL TRIAL: NCT05469607
Title: The ElectRx Study - A Neurotechnology Approach to the Treatment of IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: Florey Institute of Neuroscience and Mental Health (Unknown); University of Melbourne (Other); The Bionics Institute of Australia (Other); University of Queensland Diamantina Institute (Unknown)
Responsible Party: Principal Investigator, Dr Peter De Cruz, Head of Inflammatory Bowel Disease Unit, Austin Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HREC/52390/Austin-2019
Record Dates: First submitted 2022-07-07; First posted 2022-07-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Crohn Disease
Keywords: Resectional surgery; Post operative prevention of Crohn's recurrence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vagus Nerve Stimulator — The device consists of implantable (inside the body) and external (outside the body) components. Implantable components consist of a stimulating/recording electrode assembly that is placed around the vagus nerve in the abdomen, between the diaphragm and the stomach, a cable connecting the electrode assembly to an implantable pulse generator (IPG) that generates the stimulus and records nerve responses. The external components include a Clinical Control/Review Tool (used by the study team after implantation to adjust and periodically review the stimulation settings) and a Patient Control Unit and Charger (to turn on/off the system and perform limited adjustment of the stimulation strategy).

SUMMARY:
The purpose of this study is to evaluate the safety of vagal nerve neuromodulation in a cohort of patients operated on for Crohn's disease, in a prospective, single centre, cohort study.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older with Crohn's disease who undergo resection with an endoscopically accessible primary anastomosis which results in macroscopic normality.
* Patients having a reversal of a temporary ileostomy created after previous surgery for Crohn's disease may be enrolled provided that the reversal of the ileostomy results in a primary anastomosis and macroscopic normality of the remaining bowel.
* Patients with co-existing perianal disease may be included provided the resection has led to a primary anastomosis and macroscopic normality of the intestine.
* Patients must have proven history of Crohn's disease based on (clinical, radiologic, endoscopic and histologic criteria).

Exclusion Criteria:

* Patients with anastomosis which is endoscopically inaccessible by standard colonoscopy.
* Patients in whom there is persisting macroscopic abnormality post-surgical resection.
* Patients with Crohn's disease who have an end stoma (ileostomy or colostomy).
* Patients for whom endoscopy is not suitable due to co-morbidities or unwell clinical state
* Inability to give informed consent.
* Inability to obtain access to the anastomosis at colonoscopy.
* Suspected perforation of the gastrointestinal tract.
* Patients who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy based on endoscopic recurrence | 6 months post-operation
  Recurrence defined as the presence of any aphthous ulcers, and severe recurrence defined as an endoscopic Rutgeerts score ≥ 2 (5 aphthous ulcers or larger ulcers confined to the anastomosis)

SECONDARY OUTCOMES:
Endoscopic recurrence | 18 months post-operation
  Recurrence defined as the presence of any aphthous ulcers, and severe recurrence defined as an endoscopic Rutgeerts score ≥ 2 (5 aphthous ulcers or larger ulcers confined to the anastomosis)
Clinical recurrence | 6 months and 18 months post-operation
  Defined as recurrence of symptoms consistent with recurrent disease, necessitating new treatment, or Crohn's Disease Activity Index (CDAI) > 150
Surgical recurrence | 6 and 18 months post-operation
  Defined as the need for further intestinal surgery due to Crohn's disease

CONTACTS AND LOCATIONS:
Overall Officials: Peter De Cruz, MBBS PhD FRACP, Principal Investigator — Austin Health, Melbourne
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No